CLINICAL TRIAL: NCT05958771
Title: The Efficacy of Three Doses of Live Attenuated, Oral Rotavirus Vaccine 116E (ROTAVAC 5D) in Chilean Infants.
Brief Title: The Efficacy of Three Doses of Live Attenuated, Oral Rotavirus Vaccine 116E
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Bharat Biotech International Limited (Industry)
Responsible Party: Principal Investigator, Miguel O'Ryan Gallardo, Titular Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BBIL/Rotavac 5D-CHILE /2022
Record Dates: First submitted 2023-06-23; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Rotavirus Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Children who receive the IP (Active Comparator): The Test Article/placebo will be co-administered with the childhood vaccines that are scheduled at the regular National Program of Immunization vaccination visits around 2 months, 4 months and 6 months of age.
  Test article: ROTAVAC 5D, 3 doses. Each dose of 0.5 mL. Administered orally.
  Interventions: Drug: ROTAVAC 5D
- Children who receive placebo (Placebo Comparator): The Test Article/placebo will be co-administered with the childhood vaccines that are scheduled at the regular National Program of Immunization vaccination visits around 2 months, 4 months and 6 months of age.
  Placebo: 3 doses. Each dose of 0.5 mL. Administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ROTAVAC 5D — monovalent vaccine containing suspension of live attenuated rotavirus 116E prepared in Vero cells. Each dose contains NLT 10 e 5.0 FFU
  Arms: Children who receive the IP
Drug: Placebo — Placebo contains all the excipients of ROTAVAC 5D but without the suspension of live attenuated rotavirus
  Arms: Children who receive placebo

SUMMARY:
This is a randomized, double-blind, phase 3 study to evaluate the Efficacy, Safety, and Immunogenicity of ROTAVAC 5D, a live attenuated rotavirus vaccine in healthy infants.

A total of 5800 healthy Chilean infants will be recruited in this study and randomized to receive either vaccine or placebo in 1:1 ratio. Among these participants 300 will be categorized to immunogenicity cohort, 150 from each group, and blood samples will be collected to assess the immune response.

DETAILED DESCRIPTION:
Prior to study initiation, study clinics and offices will be set up in each of the enrollment sites. Awareness about the study will be created in the community. All categories of staff will be recruited and trained. CRFs, SOPs and registers will be developed. Regulatory and IRB approvals will be obtained. Permissions and clearances will be sought from the Government.

The study team will identify pregnant women, newborns and infants aged less than 8 weeks as potential participants. Information about the study will be shared with these families, and those willing to participate will be enrolled after obtaining consent and subsequent screening of the subject. Subjects will be enrolled in the study since 2 months + 29 days of age and will be given 3 doses of the Test Article/placebo along with childhood vaccines (which will include vaccines against diphtheria, pertussis, tetanus, Haemophilus influenzae B, Hepatitis B and IPV, and pneumococcal conjugated vaccine at 2 and 4 month of age). Participants vaccinated with a dose of vaccine from the National Immunization Program corresponding to their current age, in which more than 48 hours have passed since the last dose received, the subject will not be considered for the study. The Test Article will be liquid ORV 116E, 105.0ffu stored at 2-8°C. The Test Article/placebo will be co-administered with the childhood vaccines that are scheduled at the regular National Program of Immunization vaccination visits around 2 months, 4 months and 6 months of age. After each visit, a safety evaluation will be carried out on all participants. A card will be given to the caregivers for the daily record of temperature, diarrhea, vomiting, food refusal and/or irritability, for a period of 1 week. On day 3 and 7, the research team will contact the caregivers by telephone to note the general state of health of the infant and to collect the card. The subjects will be followed f or episodes of acute gastroenteritis every two weeks through contact by email or text message (+ 2 days), until 8 months + up to 14 days post 3 doses of vaccination. The expected duration of subjec participation is 13 months. In addition to the contacts at every two weeks follow-up, parents/primary caregiver will be advised to contact the study team whenever the subject has symptoms of gastroenteritis (GE; the operational definition of GE for this study will be the change in the habitual pattern of the stools, both in more frequent passage than is normal for the individual and/or in the decrease in stool consistency), signs or symptoms of suspected intussusception (IS, defined as stomach pain and vomiting that start suddenly and come and go several times per hour, and then later, bloody stools) or any other illness requiring hospital referral. If the caregiver report symptoms of GE, an "illness visit" will be activated. The caregiver will be asked to collect a stool specimen. The field worker will ensure that the parents/primary caregiver have stool containers available with them so that stool specimens can be collected whenever the enrolled subject has GE. In the next 24-48 hours, the stool sample will be processed with an ELISA rotavirus test. If the result is negative, the illness visit will be discontinued, and the episode will be registered. If the result is positive, a daily telephone follow-up will be carried out throughout the GE episode, up to 24 hours after the last altered stool. If during the illness visit any symptom/sign of dehydration and/or clinical severity is verified by the research team, the participant will be invited to be evaluated at the study center. During the illness visit the following variables will be collected daily by the caregiver in an illness visit card: stools number and consistency, vomiting episodes, temperature (based on subjective perception of the caregiver of potential fever, or at the same time point during the consecutive days, preferably between 2 and 8 PM), administration of ORS yes/no, number of administrations, and if possible, volume administered). If the child is hospitalized, the following information will be obtained from hospitalization charts: number and consistency of stool episodes, number of vomiting episodes, highest daily temperature, hydration evaluation, use of ORS and/or IV solutions (volume used and fluid description) duration of hospitalization, and any potential complication. If in the follow-up every two weeks of the participants, an episode that did not activate the illness visit of GE is reported or detected, the episode will be recorded and an attemp t will be made to collect as much data as possible retrospectively.

The study team will contact the parents/primary caregiver through mobile phone and collect the information of the illness visit card.

Out of the enrolled subjects, 150 from each group will constitute the "Immunogenicity Subset".

Visit 1 Baseline (vaccine at 2 Months of age + 29 days):

* The participant will be screened for eligibility based on vitals (heart rate and body temperature) and physical examination.
* If the participant is eligible (in good general health or stable preexisting disease as per the discretion of the Principal investigator).
* A study vaccine/placebo will be administered. Following vaccination, participants will remain at the study site for at least 30minutes of observation to record any immediate adverse event.
* Daily card will be given to the parent/primary caregiver.
* Blood sample (3 mL) will be collected for immunogenicity analysis in a subset of (n=300) participants prior to vaccination.

Visit 2 (vaccine at 4 Months of age, +29 days):

* Study participants will return to the OPD for vitals and physical examination (general and systemic examination). A study vaccine

  /placebo will be administered.
* Following vaccination, participants will remain at the study site for at least 30minutes of observation to record any adverse event.
* Daily card will be collected and a new card will be given to the parent/primary caregiver.

Visit 3 (vaccine at approximately 6 Months of age, +29 days):

* Study participants will return to the OPD for vitals and physical examination (general and systemic examination). A study vaccine

  /placebo will be administered.
* Following vaccination, participants will remain at the study site for at least 30minutes of observation to record any adverse event.
* Diary card will be collected and a new card will be given to the parent/primary caregiver. Visit 4 (1 Month after visit 3 ++5days): (only for immunogenicity group)
* Study participants (Subset) will return to the OPD for physical examination (general and systemic examination) and diary card will be collected.
* Blood sample (3 mL) will be collected for immunogenicity analysis in a subset of n=300.
* Diary card (Photograph) will be collected from the non-immunogenic participants. Blood samples: In the "Immunogenicity Subset", 3 ml blood specimens will be collected at baseline and 28 (+) 5 days after the third dose of the Test Article/placebo to assess the anti-rotavirus IgA antibody titer. Stool Specimens: The study team will attempt to collect a stool specimen for every GE episode, preferably within the first 2 days after episode onset . The stool specimen may be collected up to 7 days after the last day of diarrhea. The stool specimens will be sent to the laboratory. If the episode is a suspected intussusception or vaccine associated gastroenteritis that has occurred within four weeks after each dose of the Test Article/placebo, the specimen will be sent to the laboratory immediately for rotavirus testing and typing. For all ELISA RV positive samples, an aliquot of the stool specimen will be assessed for 22 enteropathogens by multiplex-PCR panel and to identify the genotype of the virus.

ELIGIBILITY:
Inclusion Criteria:

* At least one parent(s) or legally acceptable representative's consent for participation and are able to understand study procedures
* Subjects aged at least 2 months at recruitment
* No plans to move in the next 12 months

Exclusion Criteria:

* Administration of rotavirus vaccine in the past
* Participants vaccinated with a dose of vaccine from the National Immunization Program corresponding to their current age, in which more than 48 hours have passed since the last dose received
* Presence of any illness requiring hospital referral (temporary exclusion)
* Known case of immunodeficiency disease, known HIV positive
* Known case of chronic gastroenteritis disease, chronic pulmonary disease, chronic renal disease, congenital heart disease (Stable with no on-going medication).
* Any other conditions which in the judgment of the investigator warrant exclusion (e.g. no exclusion criteria but seems 'ill', investigators suspects neglect)
* Diarrhea on the day of enrollment (temporary exclusion)
* A known sensitivity or allergy to any components of the study vaccines.
* Major congenital or genetic defect.
* Has received any immunoglobulin therapy and/or blood products since birth.
* History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study, at the discretion of the principal investigator.

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5800 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subject who suffer a moderate-severe rotavirus gastroenteritis in vaccine arm as compared to placebo arm | till 8 months +14 days after administering the third dose
  Efficacy of ORV 116E in comparison to a placebo against moderate-severe rotavirus gastroenteritis defined as: episode of diarrhea (the passage of three or more loose or watery stools within a 24-hour period), with or without vomiting, that requires overnight hospitalization or rehydration therapy equivalent to World Health Organization (WHO) plan B (oral rehydration therapy) or plan C (intravenous rehydration therapy) in a medical facility such as a hospital, clinic, or supervised rural health care center

SECONDARY OUTCOMES:
Percentage of subject who suffer a severe rotavirus gastroenteritis according to the Vesikari Score in vaccine arm as compared to placebo | till 8 months +14 days after administering the third dose
  Severe rotavirus gastroenteritis: >11 on the 20 point Vesikari scoring scale, caused by non-vaccine rotavirus
Percentage of subject who suffer any severity of rotavirus gastroenteritis according to the Vesikari score in vaccine arm as compared to placebo arm | till 8 months +14 days after administering the third dose
  Any severity of gastroenteritis caused by non vaccine rotavirus
Percentage of subject who suffer moderate-severe rotavirus-only gastroenteritis (absence of co-pathogens) in vaccine arm as compared to placebo arm | till 8 months +14 days after administering the third dose
  Efficacy of ORV 116E in comparison to a placebo against rotavirus gastroenteritis defined as: episode of diarrhea (the passage of three or more loose or watery stools within a 24-hour period), with or without vomiting. Moderate-severe will be defined by the requirement of overnight hospitalization or rehydration therapy equivalent to World Health Organization (WHO) plan B (oral rehydration therapy) or plan C (intravenous rehydration therapy) in a medical facility such as a hospital, clinic, or supervised rural health care center.
  Rotavirus-only gastroenteritis will be defined as absence of co-pathogens according to Filmarray ® Gastrointestinal Panel.
Percentage of subject who suffer severe (according to Vesikari score) rotavirus-only gastroenteritis (absence of co-pathogens) in vaccine arm as compared to placebo arm | till 8 months +14 days after administering the third dose
  Efficacy of ORV 116E in comparison to a placebo against severe (>11 on the 20 point Vesikari scoring scale) rotavirus-only gastroenteritis (absence of co-pathogens according to Filmarray ® Gastrointestinal Panel )Rotavirus-only gastroenteritis will be defined as absence of co-pathogens according to Filmarray ® Gastrointestinal Panel.
Percentage of subject who suffer any severity (according to Vesikari score) of rotavirus-only gastroenteritis (absence of co-pathogens) in vaccine arm as compared to placebo arm | till 8 months +14 days after administering the third dose
  Efficacy of ORV 116E in comparison to a placebo against any severity (any score on the 20 point Vesikari scoring scale) of rotavirus only gastroenteritis (absence of co-pathogens
Percentage of subject who suffer severe (>11 on the 20 point Vesikari scoring scale) gastroenteritis irrespective of etiology in vaccine arm as compared to placebo arm | till 8 months +14 days after administering the third dose
  Efficacy of ORV 116E in comparison to a placebo against Severe (>11 on the 20 point Vesikari scoring scale) gastroenteritis irrespective of etiology
Intent to treat efficacy of ROTAVAC 5D against severe rotavirus gastroenteritis | till 8 months +14 days after administering the third dose
  Severe rotavirus gastroenteritis (≥11 on the 20 point Vesikari scoring scale) caused by non-vaccine rotavirus in the intent-to-treat population till 8 months
  +14 days after administering the third dose
Percentage of subject who suffer solicited immediate adverse events after each dose in vaccine arm as compared to placebo arm | 0 to 30 minutes after each vaccination.
  Safety of ROTAVAC 5D solicited adverse events till 30 minutes after each vaccination (immediate solicited adverse events)
Percentage of subject who suffer solicited adverse events till 7 days after each dose in vaccine arm as compared to placebo arm | 30 minutes to 7 days after each vaccination.
  Solicited adverse events occurring within 7 days after each vaccination
Percentage of subject who suffer any adverse event in the 4-week period following each dose in vaccine arm as compared to placebo arm | from day 0 to end of the study ( till 1 year (12 months) + up to 14 days)
  Unsolicited adverse events assessed from day 0 to end of the study in comparison to a placebo will be assessed in a subset of subjects Unsolicited adverse events from day 0 to 28 following each dose in comparison to a placebo will be assessed in a subset of subjects
Percentage of subject who suffer any severe adverse event during the study period in vaccine arm as compared to placebo arm | from day 0 to end of the study ( till 1 year (12 months) + up to 14 days)
  Any severe adverse event will be assessed in all subjects throughout the study period.
b. Percentage of subject who suffer intussusception during the study period in vaccine arm as compared to placebo arm | from day 0 to end of the study ( till 1 year (12 months) + up to 14 days)
  Intussusception will be assessed in all subjects throughout the study period.

OTHER OUTCOMES:
Immunogenicity rates after 3 doses of vaccine as compared to placebo arm. | 28 (+) 5 days after the third dose in comparison to baseline levels
  Immunogenicity rates after three doses of the ROTAVAC 5D in comparison to a placebo will be ascertained in approximately 150 subjects in each group assessed by four-fold rise in rotavirus-specific serum IgA antibody titers.(Time Frame: 28 (+) 5 days after the third dose in comparison to baseline levels)

CONTACTS AND LOCATIONS:
Locations (5):
- Chile (5):
  - Vacunatorio Mediped, Antofagasta, Antofagasta
  - Hospital Base de Osorno, Osorno, Los Lagos Region
  - Hospital de Puerto Montt, Port Montt, Los Lagos Region
  - Hospital Roberto del Rio, Santiago, Metropolitan Region
  - Hospital Dr. Gustavo Fricke, Viña del Mar

IPD SHARING:
Plan to Share IPD: Undecided